CLINICAL TRIAL: NCT06976749
Title: Three-Dimensional Evaluation of Pharyngeal Airway and Facial Dimension Changes in Skeletal Class II Patients Treated With Twin Block Versus Myobrace Appliances
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Lubna Makki Hussein, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1033425
Record Dates: First submitted 2025-03-19; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Class II Division 1 Adolescent Patients
Keywords: class II division 1 malocclusion; mandibular retrognathism; retrognathic mandible; Pharyngeal Airway; Twin block; Myobrace; Three-Dimensional Evaluation; facial scan
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: two-parallel arms with equal allocation ratio of 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Twin block appliance (Experimental): It consists of maxillary and mandibular appliances that fit tightly against the teeth, alveolus, and adjacent supporting structures. Adams' clasps will be used bilaterally to anchor them to the first permanent molars and lower first premolars. A short passive labial bow will be added to the upper arch and ball end clasps to the interproximal areas of the lower arch for retention. The appliance will be fabricated after a symmetric protrusive bite registration using pink modeling wax sheets, in which the patients will rehearse many times before registration. The inclined bite blocks (ramps) will be at 70 which acts as a guiding mechanism for forward displacement of the mandible. The working bite will be taken with the incisors in an edge-to-edge relationship if possible and 2 to 3 mm bite opening between the central incisors. All the subjects will be instructed to wear the appliance 24 hours/day except for brushing. If further advancement
  Interventions: Device: Twin block
- Myobrace appliance (Experimental): The appropriate size of Myobrace is chosen by using a special ruler to measure the distance between the distal portion of the lateral upper right incisor and the left, regardless of any crowding or diastema. The measure is based on the mesial-distal dimensions of the upper incisors, and not on their position. This distance is used to determine the correct size using a special table. Once chosen and inserted in patient's mouth, upper canines, even if not yet erupted, must be in their slots, so that the dental mildines coincided with the appliance's midline. In the first week, the patients will be instructed to gradually increase the wearing time of the appliance during the daytime. By the start of the second week, the patients will be instructed to wear the appliance achieving at least 8 hours during sleeping. By the end of the first 4 weeks, the patients will wear the appliances minimum of 1- 2 hours during the day plus the overnig
  Interventions: Device: myobrace appliance

INTERVENTIONS:
Device: myobrace appliance — functional appliance
  Arms: Myobrace appliance
Device: Twin block — functional appliance
  Arms: Twin block appliance

SUMMARY:
This study is intended primarily to compare the effects of two Class II correction appliances, namely Twin block and Myobrace appliances, on pharyngeal airway dimensions during the treatment of class II division 1 adolescent patients, also evaluates three dimensional (3D) changes of pharyngeal airway including: minimum cross-sectional area and volume using Cone Beam Computed Tomography (CBCT), skeletal, dentoalveolar, and soft tissue changes using cephalometric analysis, and three dimensional (3D) soft tissue changes using facial scans. The hypothesis being a consideration of no significant difference in the changes of pharyngeal airway and facial dimensions in skeletal class II patients before and after treatment with Twin block and Myobrace.

DETAILED DESCRIPTION:
This study is a multicenter randomized comparative clinical trial, employing non-stratified randomization in two-parallel arms with equal allocation ratio of 1:1. Patients will be recruited from Orthodontic Clinic at the College of Dentistry, University of Kufa, and from specialized dental centers affiliated to the Iraqi Ministry of Health, in addition to some private clinics. Initially, the patients will be assessed for eligibility to participate in the study according to the inclusion criteria. Then, the parents will be informed verbally about the purpose of the study and will be provided with the informed consent form to be signed. Patients will be treated using two types of functional appliances ( Twin Block and Myobrace) for six months. Regular follow-ups will be conducted during the course of the treatment and progress will be charted out at 4-weeks intervals.

Participants will be randomly assigned to one of two groups, each receiving one of the specified treatments over a six-month period.

Group I: Twin Block Appliance

* Design: Comprises maxillary and mandibular components anchored using Adams' clasps on the first permanent molars and lower first premolars. A passive labial bow will be incorporated into the upper arch, with ball-end clasps for additional retention.
* Bite Registration: Achieved through a symmetric protrusive bite using modeling wax, ensuring an edge-to-edge incisal relationship with a 2-3 mm bite opening between central incisors.
* Inclined Bite Blocks: Positioned at a 70° angle to facilitate forward mandibular displacement.
* Patient Instructions: Continuous wear is mandated (24 hours/day), excluding periods of oral hygiene. Adjustments using self-cured acrylic may be made for further mandibular advancement.

Group II: Myobrace Appliance

* Selection: Appropriate sizing determined by measuring the inter-canine distance using a specialized ruler.
* Fitting: Ensures alignment of upper canines within designated slots, matching the appliance's midline with the dental midline.
* Wear Protocol:
* Week 1: Gradual increase in daytime wear duration.
* Week 2 Onwards: Overnight wear targeting at least 8 hours.
* Post Week 4: Combination of 1-2 hours daytime wear plus overnight usage.
* Supplementary Activities: Incorporates exercises targeting breathing habits, tongue positioning, swallowing patterns, and lip function.

Imaging Protocols:

* Cone Beam Computed Tomography (CBCT):
* Timing: Conducted pre-treatment and at end of study .
* Positioning: Subjects seated upright with the Frankfort horizontal plane parallel to the floor, maintaining natural occlusion, relaxed lips, and resting tongue posture.
* Parameters: Scans performed using the Morita Veraview X 800 device (100 kV tube voltage, 3 mA tube current, 14 x 15 cm field of view, 0.08 mm voxel size, 18-second scan time).

three dimensional (3D) Facial Scanning:

* Equipment: Utilizes an iPhone Pro 14 equipped with the 3D Scanner App™.
* Landmark Identification: Seventeen specific facial landmarks will be marked using black eyeliner to ensure consistency.
* Participant Positioning: Subjects will be seated in a relaxed posture with a natural head position under standardized lighting conditions.
* Pre-Scan Preparations: Removal of glasses, jewelry, and use of hairbands to minimize obstructions.
* Data Processing: Captured three dimensional (3D)facial models will be exported as Standard Tessellation Language (STL) files and analyzed using Blender 3.6 LTS software for linear and angular measurements.

Data Analysis:

* three dimensional (3D) Model Reconstruction: CBCT data will be processed using ProPlan CMF 3.0 (Materialise) software.
* Segmentation: Hard tissues and upper airway structures will be delineated based on specific Hounsfield Unit (HU) thresholds.
* Pharyngeal Airway Segmentation: Divided into nasopharynx, velopharynx, glossopharynx, and hypopharynx, with precise anatomical boundaries defined for each segment.

Measurements:

* Airway Analysis: Assessment of minimum cross-sectional area, total airway volume, and pharyngeal airway length.
* Soft Tissue Evaluation: Linear and angular anthropometric measurements derived from 3D facial scans.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 10-14 years, at growth spurt phase as determined by the cervical vertebrae maturation stage (C3- C4 ) assessed by lateral cephalograms.
2. Skeletal relationship: skeletal class II (ANB angle > 4°) with normal maxilla (SNA angle 78°- 84°), and retrognathic mandible (SNB angle < 77 °).
3. Dental relationship: Moderate to severe dental class II division 1 malocclusion with overjet 6 -10 mm.
4. Convex facial profile.
5. Well aligned/mild crowding (< 4 mm) of dental arches.
6. Good to fair oral hygiene status as based on a simplified oral hygiene index (OHI-S).
7. Normal or decreased lower facial height (SN-MP angle ≤ 32).

Exclusion Criteria:

1. Previous orthodontic/orthopedic treatment.
2. Patients with dental open bite
3. Patients with obvious facial asymmetry.
4. Patients with orofacial cleft.
5. Previous extractions.
6. Presence of mandibular shifts.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
minimum cross-sectional area of the pharyngeal airway in (mm^2) using Cone Beam Computed Tomography (CBCT) | From enrollment to the end of treatment at 6 months
  3D measurements of pharyngeal airway minimum cross-sectional (mm^2) will be performed for all participants of both groups at two stages before treatment and at the end of the study using CBCT

SECONDARY OUTCOMES:
three dimensional changes in the volume of the pharyngeal airway using CBCT | From enrollment to the end of treatment at 6 months
  1. pharyngeal airway volume in (mm^3) using CBCT.
Skeletal changes using cephalometric analysis | From enrollment to the end of treatment at 6 months
  * SNA angle (relative anteroposterior position of maxilla to anterior cranial base).
  * SNB angle (relative anteroposterior position of mandible to anterior cranial base).
  * ANB angle (relative anteroposterior position of maxilla to mandible).
  * SN-Pog angle (relative anteroposterior position of chin to anterior cranial base).
  * PP-MP (Angle between palatal and mandibular plane).
  * SN-MP (Angle between SN and mandibular plane).
  * Ar-Go-Me ((Gonial Angle, it refers to the relation between the body of the mandible and the ramus).
Soft tissue changes using cephalometric analysis | From enrollment to the end of treatment at 6 months
  * NL angle (nasolabial angle).
  * U Lip-E line (upper lip to Rickett's Esthetic line).
  * L Lip-E Line (lower lip to Rickett's Esthetic line).
Dentoalveolar changes using cephalometric analysis | From enrollment to the end of treatment at 6 months
  * U1-PP (upper incisor inclination to the palatal plane).
  * L1-MP (lower incisor inclination to the mandibular plane).
Dental changes using study models | From enrollment to the end of treatment at 6 months
  overjet, overbite, inter canine, inter premolar, and inter molar widths in (mm)
three dimentional soft tissue changes using facial scans | From enrollment to the end of treatment at 6 months
  Total face height (mm) Upper anterior face height (mm) Lower anterior face height (mm) Bigonial width (mm) Mandibular length (mm) Soft tissue convexity angle Total face convexity angle Gonial angle Alar base width (mm) Lip width (mm) Nasolabial angle Labiomental angle

CONTACTS AND LOCATIONS:
Overall Officials: Lubna M Hussein, B.D.S., M.Sc. (Orthodontics), Principal Investigator — University of Baghdad
Locations (1):
- University of Baghdad, College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including 3D facial scans, CBCT airway volume measurements, and linear and angular facial measurements. The shared data will not contain any personally identifiable information. Data will be made available upon reasonable request for research purposes related to orthodontic treatment, airway evaluation, and facial growth analysis. Access will be granted to qualified researchers through a data-sharing agreement, ensuring compliance with ethical guidelines and patient privacy regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication.

REFERENCES:
- [Background] Kim SS, Kim YI, Park SB, Kim SH. Three-dimensional evaluation of the pharyngeal airway space in patients with anterior open bite. Korean J Orthod. 2023 Nov 25;53(6):358-364. doi: 10.4041/kjod22.187. Epub 2023 Jan 31. PMID 36718119
- See also: Related Info — https://e-kjo.org/journal/list.html?pn=type2